CLINICAL TRIAL: NCT07269379
Title: Intradialytic Exercise With Blood Flow Restriction by Vascular Occlusion: A New Strategy for Cardioprotection in Hemodialysis Patients
Brief Title: Intradialytic Exercise With Blood Flow Restriction in Hemodialysis Patients
Acronym: ERO-CARD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Avignon (Other)
Collaborators: Médipôle Lyon-Villeurbanne (Other); Nouvel Hôpital Civil, 1 place de l'Hôpital 67091 Strasbourg cedex (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AU-092025-CM; LAPEC/2025/ERO-CARD (Other: Avignon university)
Record Dates: First submitted 2025-11-20; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Dialysis Patients
Keywords: end stage renal disease; hemodialysis; blood flow restriction exercise; intradialytic exercise; regional myocardial function; hemorheology
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: 1. Acute phase: 3 sessions per patient, realized in a random order :
     * standard HD (HD-CONTacute)
     * HD with acute intradialytic exercise without vascular occlusion (HD-EXacute)
     * HD with acute intradialytic exercise with vascular occlusion (HD-BFREacute).
  2. Chronic phase: patients randomly assigned to one of the following 3 groups (ration 1:1:1): an exercise training program without (HD-EXChro) or with (HD-BFREChro) vascular occlusion, standard HD (HD-CONTChro) without exercise. Patients will be evaluated before and after 12 weeks of exercise rehabilitation (HD-EXChro, HD-BFREChro) or standard dialysis (HD-CONTChro).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: HD-EXChro (Experimental): Will be enrolled in a 12 weeks intradialytic exercise program without vascular occlusion
  Interventions: Other: Chronic phase - HDEX/HDBFRE; Other: Acute phase - HDEX/HDBFRE
- Experimental: HD-BFREChro (Experimental): Will be enrolled in a 12 weeks intradialytic exercise program with vascular occlusion
  Interventions: Other: Chronic phase - HDEX/HDBFRE; Other: Acute phase - HDEX/HDBFRE
- Control (No Intervention): Patients with standard HD (usual care)

INTERVENTIONS:
Other: Chronic phase - HDEX/HDBFRE — 30 min of intradialytic cycling at a moderate intensity (12-14) , starting 30min after HD onset. 3 times a week for 12 weeks. No vascular occlusion for HDEXChro. Pressure at 50% of limb occlusion pressure on both legs for HDBFREChro
  Arms: Experimental: HD-BFREChro; Experimental: HD-EXChro
Other: Acute phase - HDEX/HDBFRE — 30 min of intradialytic cycling at a moderate intensity (12-14) , starting 30min after HD onset. No vascular occlusion for HDEXacute. Pressure at 50% of limb occlusion pressure on both legs for HDBFREacute
  Arms: Experimental: HD-BFREChro; Experimental: HD-EXChro

SUMMARY:
The main objective is to evaluate in hemodialysis patients the effects of two intradialytic rehabilitation programs based on physical exercise, with or without the application of blood flow restriction, on myocardial stunning and morpho-functional cardiac remodelling, compared with usual care (i.e., dialysis without exercise). In addition, the investigators will also assess the acute effects (i.e., a single session for each condition) of physical exercise, with or without blood flow restriction, on myocardial stunning at the end of dialysis.

In comparison with a conventional exercise program, the combination of physical exercise with blood flow restriction, which synergistically and additively activates intramuscular signalling pathways related to both exercise and ischaemia, is hypothesised to result in:

1. A greater intradialytic cardioprotection, as demonstrated by a greater reduction in myocardial stunning at the end of dialysis (both in acute and chronic applications), with underlying mechanisms involving systemic and neuro-humoral pathways;
2. Significant improvements in morpho-functional cardiac remodelling, attenuation of arrhythmic disturbances, and enhancement of aerobic capacity, muscle strength, and muscle mass-effects not observed with exercise alone without blood flow restriction, considering the low exercise intensity used in the current rehabilitation program (chronic application only).

This is a three-arm randomised clinical trial with parallel groups: standard hemodialysis (HD-CONTChro), a rehabilitation program with intradialytic exercise without vascular occlusion (HD-EXChro), and a rehabilitation program with intradialytic exercise with vascular occlusion (HD-BFREChro), with a 1:1:1 allocation ratio.

To investigate the acute effects of the interventions, all patients will undergo, in a randomized order, one session of each of the three dialysis modalities-standard hemodialysis (HD-CONTacute), hemodialysis with exercise without vascular restriction (HD-EXacute), and hemodialysis with exercise with vascular restriction (HD-BFREacute)-prior to initiation of the chronic phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 20 and 79 years.
* Patients on hemodialysis for more than 3 months.
* No engagement in regular exercise outside of dialysis.
* No prior exposure to intradialytic exercise within the past six months.
* No medical contraindications to physical activity.
* Life expectancy greater than 6 months.
* Patients with relative good echogenicity

Exclusion Criteria:

* Patient is participating in another Category I interventional study, or has participated in another interventional study within the past 3 months
* The patient is in an exclusion period determined by a previous study
* The patient is under legal protection or under guardianship or curatorship It turns out to be impossible to give the patient informed information, or the patient refuses to sign the consent
* Pregnant, parturient or breastfeeding patient
* Patients with unstable coronary artery disease.
* Patients with peripheral artery disease (stage III or IV) in the lower limbs.
* Patients with limb amputation.
* Patients with musculoskeletal disorders impairing exercise.
* Presence of a pacemaker, cardiac stimulation device, or implantable cardioverter defibrillator (ICD).
* History of heart transplant.
* Patients with uncontrolled hypertension.
* Refractory anemia.
* Patients stratified as high risk for deep venous thrombosis

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2028-05-06 (Estimated); Study Completion 2028-10-06 (Estimated)

PRIMARY OUTCOMES:
Change in the number of regional wall motion abnormalities (RWMAs) | From enrollment to the end of the program at 19 weeks
  The investigators will use echocardiography to assess the number of left ventricular myocardial segments (using a 18-segment model), that demonstrate a reduction in longitudinal deformation greater than 20% at peak stress during hemodialysis, relative to baseline measurements obtained at the start of the dialysis session. Their aim is to compare the change in regional wall motion abnormalities (RWMAs) at peak stress of dialysis (i.e. 30 min before its end), in a standard HD, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  For the acute phase, the investigators will compare the number of RWMAs measured 30min before the end of each HD session between the 3 conditions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)

SECONDARY OUTCOMES:
Change in LV longitudinal strains | From enrollment to the end of the program at 19 weeks
  Using speckle tracking echocardiography, the investigators will assess variations in LV longitudinal strains during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  Strains (in %) measure the amount of myocardial longitudinal shortening of the cavity, are relatively load-independent, and can detect subclinical myocardial dysfunction, even when it is not apparent by conventional echocardiography.
  For the acute phase, the investigators will compare the changes in left ventricular (LV) longitudinal strain kinetics throughout dialysis (e.g., from the start to 30 minutes before the end of hemodialysis) among the three sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in RV longitudinal strains | From enrollment to the end of the program at 19 weeks
  Using speckle tracking echocardiography, the investigators will assess variations in RV longitudinal strains during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  Strains (in %) measure the amount of myocardial longitudinal shortening of the cavity, are relatively load-independent, and can detect subclinical myocardial dysfunction, even when it is not apparent by conventional echocardiography.
  For the acute phase, the investigators will compare the changes in right ventricular (RV) longitudinal strain kinetics throughout dialysis (e.g., from the start to 30 minutes before the end of hemodialysis) among the three sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in LA longitudinal strains | From enrollment to the end of the program at 19 weeks
  Using speckle tracking echocardiography, the investigators will assess variations in LA longitudinal strains during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  Strains (in %) measure the amount of myocardial longitudinal shortening of the cavity, are relatively load-independent, and can detect subclinical myocardial dysfunction, even when it is not apparent by conventional echocardiography.
  For the acute phase, the investigators will compare the changes in left atrial (LA) longitudinal strain kinetics throughout dialysis (e.g., from the start to 30 minutes before the end of hemodialysis) among the three sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in global constructive work | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in global constructive work during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). Global constructive work (GCW, expressed in mmHg%) will be measured using speckle-tracking echocardiography from the pressure-longitudinal strain loop generated with the dedicated module provided by the ultrasound vendor. GCW represents the work performed during shortening in systole adding negative work during lengthening in isovolumetric relaxation.
  For the acute phase, the investigators will compare the changes in LV global constructive work kinetics throughout dialysis (e.g., from the start to 30 minutes before the end of hemodialysis) among the three sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in global wasted work | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in global wasted work during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  Global wasted work (GWW, expressed in mmHg%) will be measured using speckle-tracking echocardiography from the pressure-longitudinal strain loop generated with the dedicated module provided by the ultrasound vendor. GWW represents the negative work performed during lengthening in systole adding work performed during shortening in isovolumetric relaxation.
  For the acute phase, the investigators will compare the changes in LV global wasted work kinetics throughout dialysis (e.g., from the start to 30 minutes before the end of hemodialysis) among the three sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in global work efficiency | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in global work efficiency during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). Global work efficiency (GWE, expressed in %) will be measured using speckle-tracking echocardiography from the pressure-longitudinal strain loop generated with the dedicated module provided by the ultrasound vendor. GWE will be calculated as follow: Global constructive work divided by the sum of global constructive and wasted work.
  For the acute phase, the investigators will compare the changes in LV global work efficiency kinetics throughout dialysis (e.g., from the start to 30 minutes before the end of hemodialysis) among the three sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in global myocardial work | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in global myocardial work during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  Global myocardial work (GMM, expressed in %) will be measured using speckle-tracking echocardiography from the pressure-longitudinal strain loop generated with the dedicated module provided by the ultrasound vendor. GMM represents the area of the Longitudinal strain-pressure loop.
  For the acute phase, the investigators will compare the changes in LV global myocardial work kinetics throughout dialysis (e.g., from the start to 30 minutes before the end of hemodialysis) among the three sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in left intraventricular pressure gradient | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the left intraventricular pressure gradient, measured by postprocessing color Doppler M-mode echocardiographic images during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  For the acute phase, the investigators will compare the changes in LV intraventricular pressure gradient kinetics throughout dialysis (e.g., from the start to 30 minutes before the end of hemodialysis) among the three sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in LV diameter | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in left ventricular (LV) diameter at end-systole and end-diastole, measured using Doppler M-mode echocardiography, before a standard dialysis session, before and after the 12-week program. (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
Change in LV wall thicknessess | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the LV wall thicknessess, measured by Doppler M-mode echocardiographic images before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
Change in LV volumes | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in left ventricular (LV) volumes at end-systole and end-diastole, measured using echocardiography before a standard dialysis session, before and after the 12-week program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
Change in LV mass | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the LV mass measured using echocardiography before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the LV morphology of the patients.
Change in LV global systolic function (ejection fraction) | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the LV ejection fraction measured using echocardiography before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the LV global systolic function of the patients.
Change in LV s' wave | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the LV s' wave measured by tissue Doppler imaging before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the LV regional function of the patients.
Change in LV e' wave | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the LV e' wave measured by tissue Doppler imaging before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the LV regional diastolic function of the patients.
Change in LV a' wave | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the LV a' wave measured by tissue Doppler imaging before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the LV regional diastolic function of the patients.
Change in LV E wave (global diastolic function) | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the LV E wave measured by pulsed Doppler ehocardiography during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  For the acute phase, the investigators will compare the change in LV E wave throughout the dialysis (eg before and 30min before the end of each HD) between 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute). LV E is an index of global diastolic function, characterising the LV early filling.
Change in LV A wave (global diastolic function) | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the LV A wave measured by pulsed Doppler ehocardiography during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  For the acute phase, the investigators will compare the change in LV A wave throughout the dialysis (eg before and 30min before the end of each HD) between 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute). LV A is an index of global diastolic function, characterising the LV late filling.
Change in LV E/e' | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the LV E/e' ratio measured before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the LV filling pressure of the patients.
Change in RV areas | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the RV area at end-systole and end-diastole measured before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the RV morphology and function of the patients.
Change in RV systolic function | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the RV fractional area measured using echocardiography before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the RV global systolic function of the patients.
Change in RV systolic function 2 | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the Tricuspid Annular Plane Systolic Excursion measured using echocardiography before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the RV global systolic function of the patients.
Change in RV areas | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the RV area at end-systole and end-diastole before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the RV morphology and function of the patients.
Change in RV diameter | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the RV diameter and end-systole and end-diastole, measured by Doppler M-mode echocardiographic images before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
Change in RV Et wave | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the RV Et wave by pulsed Doppler ehocardiography images before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). It will be used to characterize RV global diastolic function.
Change in RV At wave | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the RV At wave by pulsed Doppler ehocardiography images before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). It will be used to characterize RV global diastolic function.
Change in RV Et/At ratio | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the RV Et/At ratio before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). It will be used to characterize RV global diastolic function.
Change in RV e' | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the RV e' wave by tissue Doppler imaging before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). It will be used to characterize RV regional diastolic function.
Change in RV a' | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the RV a' wave by tissue Doppler imaging before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). It will be used to characterize RV regional diastolic function.
Change in RV s' | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the RV s' wave by tissue Doppler imaging before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). It will be used to characterize RV regional systolic function.
Change in tricuspid regurgitation | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the tricuspid regurgitation by continuous-wave Doppler ehocardiography before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). It will be used to characterize LV global diastolic function.
Change in RV Et/e' | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the RV Et/e' ratio before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the RV filling pressure of the patients.
Change in LA morphology and function | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in the LA volumes measured before and at end of a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the LA morphology and function of the patients.
Change in blood pressure | From enrollment to the end of the program at 19 weeks
  The investigators will measure blood pressure every 30min during a standard dialysis (i.e. from the beginning to the end of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). Their aim is to compare the changes during HD among the three groups.
  For the acute phase, the investigators will compare the change in blood pressure every 30min from the beginning to the end of HD across the three experimental conditions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in cardiac output | From enrollment to the end of the program at 19 weeks
  The investigators will measure cardiac output every 30min during a standard dialysis (i.e. from the beginning to the end of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). Their aim is to compare the changes during HD among the three groups.
  For the acute phase, the investigators will compare the change in cardiac output every 30min from the beginning to the end of HD across the three experimental conditions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in stroke volume | From enrollment to the end of the program at 19 weeks
  The investigators will measure stroke volume every 30min during a standard dialysis (i.e. from the beginning to the end of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). Their aim is to compare the changes during HD among the three groups.
  For the acute phase, the investigators will compare the change in stroke volume every 30min from the beginning to the end of HD across the three experimental conditions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in heart rate | From enrollment to the end of the program at 19 weeks
  The investigators will measure heart rate every 30min during a standard dialysis (i.e. from the beginning to the end of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). Their aim is to compare the changes during HD among the three groups.
  For the acute phase, the investigators will compare the change in heart rate every 30min from the beginning to the end of HD across the three experimental conditions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in blood level of sodium | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in blood level of sodium before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the progression of disease of the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
Change in blood level of potassium | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in blood level of potassium before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the progression of disease of the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
Change in blood level of calcium | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in blood level of calcium before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the progression of disease of the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
Change in blood level of phosphate | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in blood level of phosphate before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the progression of disease of the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
Change in blood level of vitamin D | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in blood level of vitamin D before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the progression of disease of the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
Change in blood level of parathyroid hormone | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in blood level of parathyroid hormone before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the progression of disease of the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
Change in blood level of creatinine | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in blood level of creatinine before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the progression of disease of the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
Change in creatinine clearance | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in creatinine clearance before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the progression of disease of the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
Change in blood level of urea | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in blood level of urea before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the progression of disease of the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
Change in serum level of albumin | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in serum level of albumin before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the progression of disease of the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
Change in normalized proteïn catabolic rate | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in normalized proteïn catabolic rate before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the progression of disease of the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
Change in Kt/V | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in Kt/V before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the progression of disease of the patients.
Change in serum level of c-reactive protein | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in serum level of c-reactive protein before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the progression of disease of the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
Change in complete blood count | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in complete blood count before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the blood of the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
Change in serum level of ferritin | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in serum level of ferritin before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the blood of the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
Change in transferrin saturation | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in transferrine saturation before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the blood of the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
Change in LDL cholesterol | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in LDL cholesterol before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the lipidic profile of the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
Change in HDL cholesterol | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in HDL cholesterol before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the lipidic profile of the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
Change in triglyceride level | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in triglyceride level before a standard dialysis, before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro). This will be used to characterize the lipidic profile of the patients. A blood sample will be taken directly from the arterial line of the dialysis machine at the onset of dialysis.
Change in hematocrit | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in hematocrit, measured using an hemoglobinometer, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in hematocrit kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in hemoglobin level | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in hemoglobin, measured using an hemoglobinometer, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in hemoglobin kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in interleukin-6 level | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in interleukin-6 level, measured by analyzing blood sample, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in interleukin-6 kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in interleukin-10 level | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in interleukin-10 level, measured by analyzing blood sample, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in interleukin-10 kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in tumor necrosis factor-α level | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in tumor necrosis factor-α level, measured by analyzing blood sample, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in tumor necrosis factor-α kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in ultra-sensitive c-reactive protein level | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in ultra-sensitive c-reactive protein level, measured by analyzing blood sample, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in C-reactive protein kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in intercellular adhesion molecule-1 level | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in intercellular adhesion molecule-1 level, measured by analyzing blood sample, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in intercellular adhesion molecule-1 level kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in vascular cell adhesion molecule-1 level | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in vascular cell adhesion molecule-1 level, measured by analyzing blood sample, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in vascular cell adhesion molecule-1 kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in endothelin level | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in endothelin level, measured by analyzing blood sample, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in endothelin kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in proendothelin level | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in proendothelin level, measured by analyzing blood sample, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in pro-endothelin kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in NT-pro-BNP level | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in NT-pro-BNP level, measured by analyzing blood sample, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in NT-pro-BNPkinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in BNP level | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in BNP level, measured by analyzing blood sample, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in BNP kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in cardiac troponin T level | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in cardiac troponin T level, measured by analyzing blood sample, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in cardiac troponin T kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in levels of soluble ST2 | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in levels of soluble ST2, measured by analyzing blood sample, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in soluble ST2 kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in beta2-microglobulin level | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in beta2-microglobulin level, measured by analyzing blood sample, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in beta2-microglobulin kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in indoxyl sulfate level | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in indoxyl sulfate level, measured by analyzing blood sample, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in indoxyl sulfate kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in p-Cresyl sulfate level | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in p-Cresyl sulfate level, measured by analyzing blood sample, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in p-cresyl sulfate kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in myoglobin level | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in myoglobin level, measured by analyzing blood sample, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in myoglobin kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in free light chains | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in cardiac free light chains, measured by analyzing blood sample, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in cardiac free light chain kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in whole blood viscosity | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in whole blood viscosity, measured using a cone-plate viscometer, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in whole blood viscosity kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in erythrocyte deformability | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in erythrocyte deformability, measured using an ektacytometer, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in erythrocyte deformability kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in erythrocyte aggregation | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in erythrocyte aggregation, measured using an ektacytometer, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in erythrocyte aggregation kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in fibrinogen level | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in fibrinogen level, measured by analyzing blood sample, during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in fibrinogen kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)
Change in miRNA | From enrollment to the end of the program at 19 weeks
  The investigators will assess variations in levels of circulating mi-RNAs, quantified by reverse transcription-quantitative polymerase chain reaction (RT-qPCR), during a standard dialysis (i.e. from before to the peak stress of dialysis) before and after 12 weeks of program (for HD-EXChro and HD-BFREChro) or usual care (for HD-CONTChro).
  A blood sample will be taken directly from the arterial line of the dialysis machine immediately at the onset and at the end of dialysis.
  For the acute phase, the investigators will compare the change in circulating miRNA kinetics (from the start to 30min before the end of HD) between the 3 randomized sessions (i.e. HD-CONTacute, HD-EXacute, HD-BFREacute)

CONTACTS AND LOCATIONS:
Overall Officials: Nans Florens, PhD, Principal Investigator — CHU Strasbourg
Locations (2):
- France (2):
  - CHU Strasbourg, Strasbourg
  - Medipole Lyon, Villeurbanne

IPD SHARING:
Plan to Share IPD: No